CLINICAL TRIAL: NCT01051375
Title: Examining the Effectiveness of a Wait List Intervention for the Management of Adolescent Eating Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Mark Norris, Associate Professor of Pediatrics, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09/27E
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Eating Disorders
Keywords: anorexia nervosa; bulimia nervosa; EDNOS
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Waitlist Group (Experimental): The intervention involves completion of a single workshop, provision of psychoeducational materials, and regular telephone support with a specially trained nurse-coordinator to parents of youth on our waiting list, within a month of our receiving the referral.
  Interventions: Behavioral: Psychoeducational Workshop and telephone support
- Standard of Care (No Intervention): These patients continue to receive the standard of care while awaiting formal assessment.

INTERVENTIONS:
Behavioral: Psychoeducational Workshop and telephone support — The intervention involves completion of a single workshop (delivered by a psychiatrist and adolescent health physician), provision of psycho educational materials, and regular telephone support with a specially trained nurse-coordinator to parents of youth on our waiting list.
  Arms: Waitlist Group

SUMMARY:
The current application targets patient education and enablement, implementation of best practices, continuity of care, and an improvement model to improve efficiencies by investigating whether a brief targeted intervention prior to the first formal ED assessment is efficacious in altering outcome and treatment course.

DETAILED DESCRIPTION:
The Eating Disorder Program at the Children's Hospital of Eastern Ontario (CHEO) offers a continuum of treatment options to child and adolescent patients with eating disorders (EDs). Although our own funding has increased in recent years, so too have the number of referrals, which has resulted in lengthy wait times for therapeutic assessments by our team. The current application targets patient education and enablement, implementation of best practices, continuity of care, and an improvement model to improve efficiencies by investigating whether a brief targeted intervention prior to the first formal ED assessment is efficacious in altering outcome and treatment course. It is well known that early recognition and implementation of treatment as soon as possible after the onset of symptoms is protective in eating disorders and leads to better success rates and recovery (APA Treatment Guidelines for EDs). It is hoped that the outcome of this study will influence the way in which centers look to address the ongoing issue of lengthy wait times in hopes of offering cost-effective interventions that ultimately improve patient outcomes. By offering an added level of support to families whose referral has been initiated, we hope to ease the burden of primary care providers and increase their satisfaction as it relates to patient safety concerns and complex case management.

ELIGIBILITY:
Inclusion Criteria:

* medical stability at time of referral
* completed referral to the Eating Disorders Program

Exclusion Criteria:

* patients deemed medically unstable are triaged urgently and not eligible for study inclusion

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2009-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Investigate whether a wait list intervention for patients and families who are on a wait list, improves patient presentation at the time of formal assessment, as well as 6-months post-assessment | 18 months

SECONDARY OUTCOMES:
Evaluate the impact that a wait list intervention group workshop has on caregiver knowledge, stress, and self-efficacy pertaining to eating disorders and their treatment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark Norris, MD, Principal Investigator — CHEO; Wendy Spettigue, MD, Principal Investigator — CHEO
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada